CLINICAL TRIAL: NCT04300621
Title: An Open-label, Randomized, Four-way Crossover, Single Dose Study to Investigate the Safety, Tolerability and Pharmacokinetics of Different Oral Thin Film (S)-Ketamine Formulations for Sublingual Administration in Healthy Participants
Brief Title: A Study of Different Oral Thin Film (S)-Ketamine Formulations for Sublingual Administration in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108774; 2019-004428-39 (EudraCT Number); 54135419EDI1003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-03-06; First posted 2020-03-09 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment Sequence 1: OTF 1, 4, 2, 3 (Experimental): Participants will receive a single dose of (S)-ketamine administered sublingually through OTF 1 in period 1; followed by OTF 4 in period 2; followed by OTF 2 in period 3; followed by OTF 3 in period 4, on Day 1 of each treatment period under fasted conditions. A washout period of at least 72 hours will be maintained between each treatment period.
  Interventions: Drug: OTF 1; Drug: OTF 2; Drug: OTF 3; Drug: OTF 4
- Treatment Sequence 2: OTF 2, 1, 3, 4 (Experimental): Participants will receive a single dose of (S)-ketamine administered sublingually through OTF 2 in period 1; followed by OTF 1 in period 2; followed by OTF 3 in period 3; followed by OTF 4 in period 4, on Day 1 of each treatment period under fasted conditions. A washout period of at least 72 hours will be maintained between each treatment period.
  Interventions: Drug: OTF 1; Drug: OTF 2; Drug: OTF 3; Drug: OTF 4
- Treatment Sequence 3: OTF 3, 2, 4, 1 (Experimental): Participants will receive a single dose of (S)-ketamine administered sublingually through OTF 3 in period 1; followed by OTF 2 in period 2; followed by OTF 4 in period 3; followed by OTF 1 in period 4, on Day 1 of each treatment period under fasted conditions. A washout period of at least 72 hours will be maintained between each treatment period.
  Interventions: Drug: OTF 1; Drug: OTF 2; Drug: OTF 3; Drug: OTF 4
- Treatment Sequence 4: OTF 4, 3, 1, 2 (Experimental): Participants will receive a single dose of (S)-ketamine administered sublingually through OTF 4 in period 1; followed by OTF 3 in period 2; followed by OTF 1 in period 3; followed by OTF 2 in period 4, on Day 1 of each treatment period under fasted conditions. A washout period of at least 72 hours will be maintained between each treatment period.
  Interventions: Drug: OTF 1; Drug: OTF 2; Drug: OTF 3; Drug: OTF 4

INTERVENTIONS:
Drug: OTF 1 — Participants will receive (S)-ketamine administered sublingually through OTF 1.
Drug: OTF 2 — Participants will receive (S)-ketamine administered sublingually through OTF 2.
Drug: OTF 3 — Participants will receive (S)-ketamine administered sublingually through OTF 3.
Drug: OTF 4 — Participants will receive (S)-ketamine administered sublingually through OTF 4.

SUMMARY:
The purpose of the study in healthy participants is to characterize the plasma pharmacokinetic (PK) profile of different single dose Oral Thin Film (OTF) (S)-ketamine formulations administered sublingually.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 20.0 and 28.0 kilogram per square meters (kg/m^2) inclusive (BMI=weight/height^2) with a minimum weight of 60 kilogram (kg) and a maximum of 100 kg
* Participant must be healthy based on clinical laboratory tests performed at screening. If the results of the serum chemistry panel, hematology or urinalysis are outside the normal reference ranges, retesting of an abnormal lab value(s) that may lead to exclusion will be allowed once during the screening phase
* Nonsmoker (not smoked for 3 months prior to screening)
* A woman must have a negative serum beta-human chorionic gonadotropin (beta-hCG) at screening and a negative urine pregnancy test on Day -1 of each Period
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for at least 1 month after the last study intervention administration

Exclusion Criteria:

* Cardiac arrhythmias or other cardiac disease, hematological disease, hypertension, lipid abnormalities, respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, Parkinson's disease, infection, glaucoma, epilepsy or any other illness that the Investigator considers should exclude the participant
* Positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies or human immunodeficiency virus (HIV) antibodies at screening visit
* Drinks, on average, more than 5 cups of tea/coffee/cocoa or 8 cans of cola per day
* Clinically significant acute illness within 7 days prior to each study intervention administration
* History of clinically significant drug and/or food allergies including known allergies, hypersensitivity, or intolerance to JNJ-54135419 or its excipients

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | Up to 24 hours
  Maximum plasma concentration will be reported.
Area Under the Plasma Concentration-time Curve from Time 0 To Time Of the Last Quantifiable Concentrations [AUC(0-last)] | Up to 24 hours
  Area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentrations will be reported.
Area Under the Plasma Concentration-Time Curve from Time 0 to Infinite Time [AUC(0-infinity)] | Up to 24 hours
  Area under the plasma concentration-time curve from time 0 to infinite time, calculated as the sum of AUC(last) and C(last)/lambda, in which C(last) is the last observed quantifiable concentrations will be reported.

SECONDARY OUTCOMES:
Number of Participants with Clinically Significant Abnormalities in Vital sign (Systolic Blood Pressure [SBP] and Diastolic Blood Pressure [DBP]) | Day 1
  Number of participants with clinically significant abnormalities in blood pressure (Systolic Blood Pressure [SBP], Diastolic Blood Pressure [DBP]) will be reported.
Number of Participants with Clinically Significant Abnormalities in Vital Sign (Heart Rate) | Day 1
  Number of participants with clinically significant abnormalities in vital sign (heart rate) will be reported.
Number of Participants with Clinically Significant Abnormalities in Electrocardiogram (ECGs) | Day 1 and 2
  Number of participants with clinically significant abnormalities in ECG will be reported.
Number of Participants with Clinically Significant Abnormalities in Laboratory Parameters | Day 1 and 2
  Number of participants with clinically significant abnormalities in laboratory parameters (Hematology, Clinical chemistry and routine analysis) will be reported.
Number of Participants with Adverse Events and Serious Adverse Events as a Measure of Safety and Tolerability | Up to Day 7
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- SGS Life Science Services, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency